CLINICAL TRIAL: NCT00533104
Title: Critical Limb Ischemia Treatment by Local Intra-Muscular Injection of Autologous Mononuclear Cells
Brief Title: Cell Therapy in Chronic Limb Ischemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: PIGNON / MD, Centre Hospitalier Universitaire de REIMS - FRANCE
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHRC Région 2003 / R11-05 / 95
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Peripheral Vascular Diseases
Keywords: Limb ischemia; Cell Therapy
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BM-MNC (Experimental): Patients are implanted with bone marrow - mononuclear cells
  Interventions: Procedure: BM-MNC preparation
- PB-MNC (Experimental): Patients are implanted with peripheral blood - mononuclear cells
  Interventions: Procedure: PB-MNC preparation

INTERVENTIONS:
Procedure: BM-MNC preparation — For autologous bone marrow - mononuclear cells preparation, 500ml of bone marrow are collected under general anaesthesia; mononuclear cells are separated using a blood-cells separator (COBE SPECTRA, GAMBRO BCT) and concentrated to produce a final volume of 40ml.
  Cells are implanted 1 to 3 hours after preparation by multiple intramuscular injections into the gastrocnemius of the ischemic leg.(30 injection sites, 1 to 1.5 cm deep, spaced 1 cm apart,1 ml per injection).
  Arms: BM-MNC
Procedure: PB-MNC preparation — Peripheral blood - mononuclear cells are collected through cytapheresis with the same blood-cells separator which is adjusted to obtain a 40 mL cell product. No previous mobilization with hematopoïetic growth-factor is administered.
  Cells are implanted 1 to 3 hours after preparation by multiple intramuscular injections into the gastrocnemius of the ischemic leg.(30 injection sites, 1 to 1.5 cm deep, spaced 1 cm apart,1 ml per injection).
  Arms: PB-MNC

SUMMARY:
The primary focus of the trial is safety and efficacy of the intra-muscular implantation of either bone-marrow, or peripheral blood mononuclear cells, in critical limb ischemia, as judged by the proportion of patients which are alive without major amputation 6 months after inclusion.

DETAILED DESCRIPTION:
Critical limb ischemia is a frequent situation whose incidence can be evaluated to 500 to 1,000 per million per year. Limb salvage is the main goal of therapy and is usually attempted by surgical or percutaneous vascularization procedures. However approximately 25 % of patients are not suitable for such procedures and it was estimated that less than half of these patients were alive without any major amputation after 6 months. In this setting cell therapy has been proposed to stimulate angiogenesis. The first significant experience in humans was reported by TATEISHI-YUYAMA et al who showed that autologous implantation of bone marrow mononuclear cells (BM-MNC) was safe and increased blood flow in ischemic limbs resulting in clinical improvement. The same authors did not observe any efficacy of peripheral blood mononuclear cells (PB-MNC). Subsequently other publications reported positive effects of PB-MNC which were harvested after previous treatment with haematopoietic growth factor to induce a mobilization of stem cells. However such a treatment could have deleterious effects in patients presenting with advanced arterial disease. In this context we propose a prospective bi-centric trial to evaluate the safety and efficacy of autologous implantation of either BM-MNC or PB-MNC without previous mobilization with hematopoïetic factor, in patients with critical limb ischemia.

The trial is designed in two steps : a first series of eight patients are treated with BM-MNC and the following eight will receive PB-MNC. An interim analysis is planned after these first sixteen cases. Based on this analysis, it will be decided to include 12 further patients with each type of cells.Patients are consecutively included as soon as they present with appropriate criteria and are not selected to receive one or another type of cells.

Before implantation, MNC counts, differential and viability are determined. CD34+, CD34+/CD133+ and CD34+/CD133+/flk-1+ cells are counted by flow-cytometry.

Clinical symptoms and TcPO2 are monitored 1, 2, 7 and 14 days, 1, 3, and 6 months after cell implantation. Blood cell count, C-reactive protein, Interleukin-6, tumor necrosis factor-α, myoglobin, and creatinin-kinase are determined at day 0, 1, 3 and 7 ; blood vascular-endothelial-growth-factor (VEGF) level and CD34+, CD34+/CD133+ blood cells are measured before and 72 hours after implantation

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral critical chronic limb ischemia but not suitable candidates for non-surgical or surgical revascularization
* Before being included, the patient must be screened for human immunodeficiency virus, hepatitis B virus, hepatitis C virus, treponema pallidum

Exclusion Criteria:

* Buerger disease
* Ischemic ulcers with infectious symptoms
* Diabetes mellitus with HbA1c > 7,5% or with proliferative retinopathy
* Past or current malignancy
* Contra-indication to general anaesthesia
* Chronic haemodialysis
* Prothrombin Time < 60%,
* Recent onset (within 3 months) of myocardial infarction or brain infarction
* Coronary angioplasty within 1 year
* Atrial fibrillation, mechanical mitral prosthetic valve
* Unexplained hematological abnormality.
* Expected life span less than six months
* Patient not competent to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Survival without major amputation | 6 months after implantation

SECONDARY OUTCOMES:
clinical symptoms and haemodynamic parameters | Within 6 months after implantation

CONTACTS AND LOCATIONS:
Overall Officials: Bernard PIGNON, MD, Study Director — University Hospital REIMS FRANCE; Marie-Antoinette SEVESTRE, MD, Principal Investigator — University Hospital AMIENS FRANCE
Locations (1):
- Patricia LEMARCHAND, Nantes, France

REFERENCES:
- [Result] Pignon B, Sevestre MA, Chatelain D, Albertini JN, Sevestre H. Histological changes after implantation of autologous bone marrow mononuclear cells for chronic critical limb ischemia. Bone Marrow Transplant. 2007 May;39(10):647-8. doi: 10.1038/sj.bmt.1705656. Epub 2007 Mar 26. No abstract available. PMID 17384655
- [Derived] Al-Rifai R, Nguyen P, Bouland N, Terryn C, Kanagaratnam L, Poitevin G, Francois C, Boisson-Vidal C, Sevestre MA, Tournois C. In vivo efficacy of endothelial growth medium stimulated mesenchymal stem cells derived from patients with critical limb ischemia. J Transl Med. 2019 Aug 9;17(1):261. doi: 10.1186/s12967-019-2003-3. PMID 31399109
- [Derived] Capiod JC, Tournois C, Vitry F, Sevestre MA, Daliphard S, Reix T, Nguyen P, Lefrere JJ, Pignon B. Characterization and comparison of bone marrow and peripheral blood mononuclear cells used for cellular therapy in critical leg ischaemia: towards a new cellular product. Vox Sang. 2009 Apr;96(3):256-65. doi: 10.1111/j.1423-0410.2008.01138.x. Epub 2008 Dec 15. PMID 19207166